CLINICAL TRIAL: NCT05138393
Title: PREventing Mild Idiopathic SCOliosis PROgression (PREMISCOPRO): a Randomized Controlled Trial Comparing Scoliosis-specific Exercises to Observation in Mild Idiopathic Scoliosis
Brief Title: Scoliosis-specific Exercises for Mild Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Paul Gerdhem, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ED-PG-AA-2021-SSE
Record Dates: First submitted 2021-11-05; First posted 2021-12-01 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Scoliosis
Keywords: Idiopathic scoliosis; Randomized controlled trial; Exercise; Rehabilitation; Self-correction
MeSH Terms: conditions — Motor Activity | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active self-corrective exercises (Experimental): An active self-correction tailored to the individual type of curve and clinical presentation will be applied with the aim to correct the scoliosis in all three planes. Patients will also be informed and educated in task oriented activities of daily living. Training goals are directed towards postural control, spinal stability, muscular stabilization and endurance in corrective postures. Patients will have outpatient sessions once every two weeks the first 3 months and perform the exercises at home in 30-minutes sessions three times per week. Patients are encouraged to continue with non-specific self-mediated physical activities of moderate intensity at least 60 minutes daily. Compliance will be monitored through a mobile application (Physitrack) where the patients record their sessions and can have contact with the research personnel. A cognitive behavioral therapy approach to reinforce physical activity will be performed every 6 months.
  Interventions: Other: Active self-corrective exercises
- Observation (Active Comparator): Patients are encouraged to continue with non-specific self-mediated physical activities of moderate intensity at least 60 minutes daily, for the entirety of the study. A cognitive behavioral therapy approach to reinforce physical activity will be performed every 6 months.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Active self-corrective exercises — Scoliosis specific exercises with an Active self-corrective approach. Non-specific physical activity 60 minutes per day.
  Arms: Active self-corrective exercises
Other: Observation — Non-specific physical activity 60 minutes per day.
  Arms: Observation

SUMMARY:
Idiopathic scoliosis is the most common spinal deformity in children and adolescents with an estimated prevalence of 3%. About one tenth of the children with scoliosis develop a deformity that requires treatment with brace or surgery with the current treatment protocol. In Sweden, mild scoliosis curves not requiring treatment, but at risk for progression during childhood, are only observed until skeletal maturity without active treatment. If progression occurs and treatment is required, standard treatment consists of bracing 20 hours or more per day. Scoliosis-specific exercises have been reported to be a possible treatment modality in terms of halting progression in mild scoliosis, but the findings are not generally accepted.

DETAILED DESCRIPTION:
Mild forms of idiopathic scoliosis are usually observed with regular clinical and radiological follow-ups during growth periods. Scoliosis specific exercises have been used as a method aiming to halt progression and ultimately avoid the need of brace treatment. However, many cases of mild idiopathic scoliosis will not progress irrespective of treatment. As of today, there are a number of different methods and approaches to scoliosis specific exercises, but all with the aim to correct scoliosis in the sagittal, frontal and transverse plane.

In a multicenter randomized controlled trial, the investigators seek to compare an active self corrective management of scoliosis specific exercises to observation for patients with mild scoliosis. Skeletally immature patients with mild idiopathic scoliosis will be randomized in an online module through the Swedish spine register (www.swespine.se), to receive either the intervention or observation. Outcome assessors will be blinded for the type of management the patients are having. Compliance will be monitored with a mobile application (Physitrack) where the patients and their families can have direct access to the research personnel and their treatment. Outcome measures include changes in curve severity, quality of life, number of patients requiring brace treatment and clinical outcomes. All patients will be evaluated with clinical follow-ups every six months and both clinical and radiological follow-ups each twelve months until either progression occurs or skeletal maturity is reached. Individuals progressing and requiring brace treatment will be offered standard TLSO or nighttime brace to be worn 20 hours and 8 hours, respectively, per day and will be followed in the same way as other participants. Skeletal maturity is defined as less than 1 cm of growth in six months. All patients will be encouraged to be physically active for 60 minutes per day. When skeletal maturity has occured, patients will have clinical and radiological follow-ups at 2, 5 and 10 years after treatment termination. Based on a hypothesized failure rate of 10% in the scoliosis specific exercise group and 39% in the observation group, with a significance level of 5% and a power of 80% and consideration for dropout of up to 20% and an additional adding of five individuals per group, an estimated number of 45 individuals in each group is required.

For individuals who are not willing to be randomized and participate in the study, observation will be offered and these individuals will serve as an observational group with similar follow-ups and will be asked to answer the same survey as the study groups will do.

ELIGIBILITY:
Inclusion Criteria:

* Cobb 15-24 degrees
* Skeletally immature, Sanders score of 4 or less and Risser < 2.
* No menarche for females
* Aged 9-15 years
* Apex of the primary curve at T7 or caudal

Exclusion Criteria:

* Non-idiopathic scoliosis (i.e. neuromuscular, syndromic or congenital scoliosis)
* No previous surgical or brace treatment for scoliosis

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2037-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients progressing in curve severity | Measured at each radiological (annual) follow-up until skeletal maturity. Skeletal maturity is defined as less than 1 cm body height increase in 6 months
  Increase in curve severity (Cobb angle) of more than 6 degrees on two consecutive full-spine frontal radiographs as compared with baseline

SECONDARY OUTCOMES:
Angle of trunk rotation | At each six-month follow-up and at 2, 5, 10 years after skeletal maturity
  Angle of trunk rotation in forward bending, assessed according to Adams forward bending test with Bunnell's scoliometer
Patient-reported outcome measures | At each six-months follow-up and 2, 5, 10 years after skeletal maturity
  Scoliosis Research Society-22r questionnaire (SRS-22r) ranging from 1 (worst) to 5 (best)
Patient-reported outcome measures | At each six-month follow-up and 2, 5, 10 years after skeletal maturity
  The child-friendly EQ-5D version (EQ-5D-Y) with values ranging from 1 (best) to 3 (worst)
Patient-reported outcome measures | At each six-month follow-up, and 2, 5, 10 years after skeletal maturity
  Pictorial part of Spinal Appearance Questionnaire (pSAQ) with values ranging from 7 (best) to 35 (worst)
Patient-reported outcome measures | At each six-month follow-up, and 2, 5, 10 years after skeletal maturity
  International Physical Activity Questionnaire-short form (IPAQ-SF) where data will be presented as energy expenditure, Metabolic Equivalent Task (MET) minutes, and proportion of individuals reaching moderate activity level. Moderate activity level is considered if 3 or more days of vigorous activity of at least 20 minutes per day, 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day, or 5 or more days of any combination of walking, moderate-intensity, or vigorous-intensity activities accumulating at least 600 MET-minutes per week
Brace treatment | At each six-months follow-up and 2, 5, 10 years after skeletal maturity
  Number of patients needing brace treatment. Indication for brace treatment is progression of more than 6 degrees on standing frontal radiograph and a primary curve surpassing 25 degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Diarbakerli, PT, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Linköping university hospital, Linköping
  - Karolinska university hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
IPD underlying published manuscripts will be accessible for other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol will be submitted to a peer-reviewed journal.
Access Criteria: The investigators in charge will be responsible for reviewing access requests. Crude data, randomization procedures and intervention details can be shared with other researchers upon request.